CLINICAL TRIAL: NCT02092948
Title: A Phase I Open Label Study to Evaluate the Tumor-targeting Properties and Safety of 124I-A11 PSCA Minibody in Patients With Metastatic Prostate, Bladder and Pancreatic Cancer.
Brief Title: Phase I Study to evaluate124I-A11 PSCA Minibody in Patients With Metastatic Prostate, Bladder and Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: ImaginAb, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-000922; MNBD-PROT01 (Other: Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2016-05

CONDITIONS: Prostate Cancer; Pancreatic Cancer; Bladder Cancer
Keywords: metastatic; PSCA; minibody; PET/CT
MeSH Terms: conditions — Prostatic Neoplasms; Pancreatic Neoplasms; Urinary Bladder Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental): Patients will receive one intravenous dose of 4 mg, 20mg or 40 mg of A11 minibody labeled with 5 mCi (185 MBq) of 124I, followed by [124I] PSCA-Minibody PET/CT imaging of the whole body.
  Interventions: Radiation: [124I] PSCA-Minibody PET/CT imaging of the whole body

INTERVENTIONS:
Radiation: [124I] PSCA-Minibody PET/CT imaging of the whole body — Whole body Imaging

SUMMARY:
The purpose of the study is to determine whether positron emission tomography (PET), using the new imaging drug [124 I] PSCA-Minibody can be used for imaging prostate, pancreatic or bladder cancer that has spread to the bones and soft tissues (e.g., lymph nodes, lungs, etc.). The PET imaging drug tested in this study binds to the cell marker called Prostate Stem Cell Antigen (PSCA), which is present on certain prostate, pancreatic and bladder cancers.

DETAILED DESCRIPTION:
The people doing this study want to find out:

1. Can the [124 I] PSCA-Minibody be used to image prostate, pancreatic and bladder cancer?
2. How much of the PSCA Minibody needs to be used to see the prostate, pancreatic or bladder cancer?
3. Does the PSCA Minibody see more/same/fewer lesions than are identified on traditional scans such as bone scan or CT scan?

To answer these questions, we want to evaluate how [124 I] PSCA-Minibody is distributed throughout the body in 20 patients with prostate, pancreatic or bladder cancer. This is done with PET/CT imaging. A PET/CT scan is a non-invasive x-ray test that uses a special camera to take pictures of the inside of your body. It can "see" the radiation given off by tiny particles called positrons in the radioactive drug injected into you while also taking pictures of the organs within the body. For this study the radioactive substance is [124 I] PSCA-Minibody.

The scanning for this study is done with an imaging procedure in the department of Nuclear Medicine during which the experimental drug [124 I] PSCA-Minibody will be administered by intravenous (i.v.) infusion. An experimental drug is one that is not yet approved by the US Food and Drug Administration (FDA). [124 I] PSCA-Minibody is a combination of a monoclonal antibody, and I-124, a radioactive type of iodine. The iodine will make the antibody and the cancer cells visible in a PET scan. PET stands for positron emission tomography and uses radioactivity to image the inside of the body. A CT scan uses x-rays to look at the internal organs in the body. This study will use a combination PET/CT to look at the cancer cells in your body that have taken up the study agent as well as to see their location in your body.

ELIGIBILITY:
Inclusion Criteria (subjects must meet all of the following criteria in order to be enrolled in this study):

1. Histological diagnosis of prostate, bladder or pancreatic cancer.
2. Evidence of recurrent metastatic disease demonstrated by an abnormal bone scan, CT scan or MRI, or FDG-PET within 6 weeks (with no new interval treatment before imaging trial)
3. Expected survival ≤ 6 months
4. Provide written informed consent and willing to comply with protocol requirement
5. ≥ 18 years of age
6. The following laboratory results should be within the following limits within 4 weeks prior to study day 1:

   1. PSA > 5 (only for prostate cancer patients)
   2. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/l
   3. Platelet count ≥ 100 x 10^9/l
   4. Serum bilirubin ≤ 2.0 mg/dl
   5. Aspartate amino transaminase (AST) ≤ 2.5 x ULN
   6. Alanine aminotransferase (ALT) ≤ 2.5 x ULN
   7. Serum creatinine ≤ 2.0 mg/dl (calculated creatinine clearance > 45 ml/min)
7. Able to undergo imaging studies, as well as conventional bone and body imaging, as well as 124I-A11 PSCA minibody experimental scan.

Exclusion Criteria (subjects meeting any of the following criteria will not be enrolled in this study):

1. Inadequate venous access (two antecubital or equivalent venous access sites)
2. Administration of a radionuclide within 5 physical half-lives prior to projected administration of 124I-A11 PSCA minibody
3. New York Heart Association Class III/IV cardiac disease.
4. History of autoimmune hepatitis
5. Treatment with any experimental therapy within 30 days prior to enrollment or current participation in any other interventional clinical study
6. Subjects weighing ≥ 350 lbs or are unable to fit in the imaging gantry
7. Any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete good quality data.
8. Iodine Allergy, hyperthyroidism, or Grave's disease.
9. Any other disease or medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-08-22 (Actual); Primary Completion 2017-01-06 (Actual); Study Completion 2017-01-06 (Actual)

PRIMARY OUTCOMES:
Assess the safety of [124I] PSCA-Minibody | up to 3 months
  Safety measures: adverse events including laboratory adverse events will be graded and summarized according to the National Cancer Institute CTCAE, version 4.03.
  * Laboratory tests (CBC with differential, platelets, serum electrolytes, BUN, creatinine, chemistry, urine analysis)
  * Vital signs (upright and supine blood pressure, heart rate, respiratory rate, oral temperature, and weight)
  * Physical examination
  * HAMBA tier in serum

SECONDARY OUTCOMES:
Assess the ability of [124I] PSCA-Minibody to image known metastatic disease | 1 Day of scan
  Binary qualitative reading of [124I] PSCA-Minibody based PET imaging in subjects with known metastatic prostate, pancreatic, or bladder cancer to decide on the presence or absence of targeting to this cancer.
Compare the sensitivity and specificity of [124I] PSCA-Minibody with conventional imaging | 1 Day of scan
  Number, localization and size of metastatic lesions by 124I-A11 based PET/CT imaging and comparison to standard of care imaging with CT and bone scan.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Pantuck, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States